CLINICAL TRIAL: NCT01959425
Title: Safety of Oral Anticoagulation Therapy Withdrawal After Successful Cardiac Ablation in Patients With Atrial Fibrillation and Associated High Risk Factors for Embolic Events (OAT Pilot Study)
Brief Title: Oral Anticoagulation Therapy Pilot Study
Acronym: OAT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OAT-149
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Results first posted 2020-12-17 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Anticoagulation; Oral; Paroxysmal atrial fibrillation; Patients post successful cardiac ablation; Symptomatic high-burden paroxysmal AF; 3 months post procedure; Remain free from AF recurrence
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Off OAT Group (Test) (Experimental): Discontinuation of OAT Therapy
  Interventions: Other: Off OAT Group (Test)
- On OAT Group (Control) (Other): Continuation of OAT Therapy
  Interventions: Other: On OAT Group (Control)

INTERVENTIONS:
Other: Off OAT Group (Test) — Discontinuation of OAT Therapy
  Arms: Off OAT Group (Test)
Other: On OAT Group (Control) — Continuation of OAT Therapy
  Arms: On OAT Group (Control)

SUMMARY:
The objective of this study is to determine the safety of discontinuing oral anticoagulation therapy in high risk patients who have had a successful cardiac ablation and remain AF recurrence free for 3 months post ablation.

DETAILED DESCRIPTION:
Patients undergoing successful cardiac ablation for atrial fibrillation who remain AF recurrence-free 3 months after successful ablation and continue to meet the inclusion/exclusion criteria will be screened for enrollment in the trial. After fulfilling all of the inclusion/exclusion criteria, patients who consent to participate in the study and remain AF recurrence-free will be randomized to one of two study arms: (1) OAT Withdrawal (Test) Group or (2) OAT (Control) Group and participate in the Evaluation Period (12 months).

ELIGIBILITY:
Inclusion Criteria:

1. Successful cardiac ablation for AF
2. Documented freedom from AF recurrence (symptomatic or asymptomatic arrhythmic recurrences lasting longer than 30 seconds) 3 months after successful cardiac ablation (AF recurrence during 3-month blanking period is excluded).
3. Patient must have been on a commercially approved anticoagulation therapy for at least two (2) months prior to randomization in the OAT Study.
4. CHADS2 score ≥ 2 or CHA2DS2-VASc score (≥3)
5. Left ventricular ejection fraction > 25%
6. LA size < 65
7. High risk for thromboembolic events (i.e., CHADS2 score ≥ 2 or CHA2DS2-VASc score ≥ 3) and require OAT before undergoing cardiac ablation
8. Able and willing to comply with all pre- and follow-up testing and requirements
9. Signed informed consent form
10. Age 18 years or older

Exclusion Criteria:

1. OAT required for reasons not related to AF (i.e., prosthetic valve, PV stenosis, previous pulmonary embolism, presence of spontaneous echo contrast [SEC] at standard echo performed at 3-months follow-up).
2. Any cardiac surgery within the past 60 days (2 months) or valvular cardiac surgical procedure at any time (i.e., ventriculotomy, atriotomy, and valve repair or replacement and presence of a prosthetic valve)
3. Previous myocardial infarction (MI) or a percutaneous coronary intervention PCI within the past 3 months
4. Awaiting cardiac transplantation or other cardiac surgery within the next 365 days (12 months)
5. Documented left atrial thrombus
6. Significant pulmonary disease, (e.g., restrictive pulmonary disease, constrictive or COPD) or any other disease or malfunction of the lungs or respiratory system that produces chronic symptoms
7. Significant medical problem that in the opinion of the investigator would preclude enrollment in this study
8. Women who are pregnant (as evidenced by pregnancy test if pre-menopausal)
9. Acute illness or active systemic infection or sepsis
10. Unstable angina
11. Contraindication to anticoagulation (i.e., heparin, warfarin or another commercially available anticoagulation medication)
12. History of blood clotting or bleeding abnormalities
13. Life expectancy less than 360 days (12 months)
14. Uncontrolled Heart Failure or NYHA Class III or IV heart failure
15. Enrollment in a clinical study evaluating another device or drug, within the past 6 months
16. Unable or unwilling to comply with protocol requirements

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-04-17 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2019-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, MD, Principal Investigator — Texas Cardiac Arrhythmia Research Foundation; Antonio Raviele, MD, Principal Investigator — Dell'Angelo Hospital; Michael Riley, MD, Principal Investigator — University of Pennsylvania; Karl Heinz Kuck, MD, Principal Investigator — Hanseatisches Herzzentrum, Asklepios Klinik; Michel Haissaguerre, MD, Principal Investigator — Hospital Cardiologigue du Haut-Leveque; Pierre Jais, MD, Principal Investigator — Hospital Cardiologigue du Haut-Leveque; Sakis Themistoclakis, MD, Principal Investigator — Dell'Angelo Hospital

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled April 17, 2013. The last subject was enrolled January 25, 2019.
Pre-assignment Details: This was a prospective, multicenter, randomized, controlled, two arm, 1:1 design. Enrolled subjects N=80 (subjects signed informed consent). 63 subjects underwent study procedures, 17 subjects were excluded prior to randomization. According to protocol, enrolled subjects = subjects who sign the study's informed consent form.
Period: Overall Study
Arm/Group | Off OAT Group (Test) | On OAT Group (Control)
Started | 32 | 31
Completed | 20 | 23
Not Completed | 12 | 8
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Discontinued Subjects | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Off OAT Group (Test) | On OAT Group (Control) | Total
Number analyzed (Participants) | 32 | 31 | 63
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.7 (5.85) | 66.0 (11.09) | 66.9 (8.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 21 | 21 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 27 | 25 | 52
  Unknown or Not Reported | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 0 | 1
  White | 24 | 28 | 52
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Occurrence of Any Major Thromboembolic Event
Description: Composite endpoint represented by the occurrence of any major thromboembolic event (stroke [i.e., ischemic, hemorrhagic or cryptogenic] that is an acute onset of a focal neurologic deficit of presumed vascular origin lasting for ≥24 hours or resulting in death) or major hemorrhagic complication (major bleeding) during the 12-month Evaluation Period.
Time Frame: 12 months
Measure: Number; unit: Number of Participants
Arm/Group | Off OAT Group (Test) | On OAT Group (Control)
Number analyzed (Participants) | 32 | 31
Number of Participants | 0 | 0

2. Secondary Outcome: Percentage of Participants With Minor Bleeds
Description: Any clinical bleed that does not meet criteria for a major hemorrhagic event during the 12-month Evaluation Period.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Off OAT Group (Test) | On OAT Group (Control)
Number analyzed (Participants) | 32 | 31
Percentage of Participants | 0 [0 to 0] | 3.2 [0.1 to 16.7]

3. Secondary Outcome: Percentage of Participants Hospitalized With Any Thromboembolic or Major Hemorrhagic Event
Description: Hospitalization due to any thromboembolic or major hemorrhagic event during the 12-month Evaluation Period.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Off OAT Group (Test) | On OAT Group (Control)
Number analyzed (Participants) | 32 | 31
Percentage of Participants | 3.1 [0.1 to 16.2] | 0 [0 to 0]

4. Secondary Outcome: Percentage of Expired Participants
Description: All cause mortality during the 12-month Evaluation Period.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Off OAT Group (Test) | On OAT Group (Control)
Number analyzed (Participants) | 32 | 31
Percentage of Participants | 0 [0 to 0] | 0 [0 to 0]

5. Secondary Outcome: Mean SF-36 Quality of Life Scores of Participants at Baseline, 3 Months, and 12 Months: Physical Component Summary (PCS)
Description: The 36-Item Short Form Health Survey (SF-36) is a validated health-related quality of life (HRQOL) tool used to measure the physical and mental health status of the study population. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 score on the assumption that each question carries equal weight. Scores can be summed together to contribute to two summary scores, a physical component score and a mental component score. The lower the score, the more disability.
Time Frame: Baseline, 3 months, 12 months
Population: The number of participants analyzed at each time point reflects the number of surveys collected at that time point for each group. Participants may have refused to complete the survey, or were exited from the study prior to the visit.
Measure: Mean (Standard Deviation); unit: Points on SF-36 scale
Arm/Group | Off OAT Group (Test) | On OAT Group (Control)
Number analyzed (Participants) | 32 | 31
Points on SF-36 scale
  Mean Score at Baseline: number analyzed (Participants) | 31 | 30
  Mean Score at Baseline | 49.8 (8.56) | 50.0 (8.24)
  Mean Score at 3 Months: number analyzed (Participants) | 28 | 26
  Mean Score at 3 Months | 52.3 (6.85) | 50.3 (8.66)
  Mean Score at 12 Months: number analyzed (Participants) | 19 | 21
  Mean Score at 12 Months | 49.3 (8.60) | 50.0 (7.06)

6. Secondary Outcome: Mean SF-36 Quality of Life Scores of Participants at Baseline, 3 Months, and 12 Months: Mental Component Summary (MCS)
Description: as for outcome 5
Time Frame: Baseline, 3 months, 12 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Points on SF-36 scale
Arm/Group | Off OAT Group (Test) | On OAT Group (Control)
Number analyzed (Participants) | 32 | 31
Points on SF-36 scale
  Mean Score at Baseline: number analyzed (Participants) | 31 | 30
  Mean Score at Baseline | 51.5 (8.33) | 54.8 (8.53)
  Mean Score at 3 Months: number analyzed (Participants) | 28 | 26
  Mean Score at 3 Months | 52.8 (9.94) | 53.7 (10.47)
  Mean Score at 12 Months: number analyzed (Participants) | 19 | 21
  Mean Score at 12 Months | 53.2 (8.70) | 53.5 (9.79)

7. Secondary Outcome: Percentage of Participants With Atrial Fibrillation Recurrence
Description: Recurrence of atrial fibrillation during the 12-month Evaluation Period. Subjects with recurrence of atrial fibrillation were immediately exited from the study.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Off OAT Group (Test) | On OAT Group (Control)
Number analyzed (Participants) | 32 | 31
Percentage of Participants | 18.8 [7.2 to 36.4] | 12.9 [3.6 to 29.8]

8. Secondary Outcome: Percentage of Participants With Repeat Ablation
Description: Repeat ablations performed due to recurrence of atrial fibrillation during the 12-month Evaluation Period. Subjects that required a repeat ablation were immediately exited from the study.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Off OAT Group (Test) | On OAT Group (Control)
Number analyzed (Participants) | 32 | 31
Percentage of Participants | 0 [0 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: 12 Months
Arm/Group | Off OAT Group (Test) | On OAT Group (Control)
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/31
Serious Adverse Events (participants affected / at risk) | 6/32 | 2/31
Other Adverse Events (participants affected / at risk) | 0/32 | 4/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Off OAT Group (Test) (N=32) | On OAT Group (Control) (N=31)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Arterial bypass thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Off OAT Group (Test) (N=32) | On OAT Group (Control) (N=31)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Joint Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any results communications proposed to be published or presented shall be submitted to Sponsor at least 60 days prior to public release to permit Sponsor to direct removal of any confidential information contained therein. The first results communications should be a multicenter, joint publication. If a multicenter publication is not submitted by the Sponsor or designee within 12 months of the Study conclusion, PIs may publish results from their institution in accordance with the above.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-10-21): https://cdn.clinicaltrials.gov/large-docs/25/NCT01959425/Prot_SAP_000.pdf